CLINICAL TRIAL: NCT04026373
Title: RAC Pilot - The Feasibility and Effectiveness of a Brief Preventive Intervention Following Psychological Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sadie Larsen, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00024745
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Prolonged Exposure (Experimental)
  Interventions: Behavioral: modified Prolonged Exposure
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: modified Prolonged Exposure
  Arms: modified Prolonged Exposure
Behavioral: Treatment as usual — May include consult to health psychology and any follow-up deemed appropriate
  Arms: Treatment as usual

SUMMARY:
The investigators proposed to compare a modified Prolonged Exposure intervention to treatment as usual within a hospitalized injured trauma survivor sample, to determine with this intervention could prevent the development of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive motor vehicle crash (MVC), industrial accident, and physical assault trauma survivors (i.e. victims of gunshot wounds, stab wounds), ages 18-75, to include both men and women, without evidence of serious cognitive impairment, admitted to the trauma surgery service at Froedtert Hospital beginning at the start of the funding period will be considered for recruitment.

Exclusion Criteria:

* Individuals who:

  1. have evidence of moderate to severe cognitive impairment secondary to trauma-related head injury,
  2. have self-inflicted injury,
  3. are more than 2 weeks post-trauma,
  4. do not meet the DSM-5 definition of a traumatic stressor for PTSD,
  5. screen positive for a current substance abuse problem ((i.e. intoxication and memory loss upon arrival or a current substance use diagnosis),
  6. are non-English speaking,
  7. are not medically stable,
  8. cannot identify a support person to attend a session with them
  9. do not score a 2 or more on the 5-item PTSD subscale of the 9-item screen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale | Three months post-trauma
  Total score will be examined. Range is 0 to 80, with higher scores indicating higher severity of PTSD symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen SE, Hunt JC, Geier T, Heyrman K, Schumann N, Brandolino A, Timmer-Murillo S, Bergner C, Larson C, deRoon-Cassini TA. A Randomized Trial of Modified Prolonged Exposure to Prevent the Development of Posttraumatic Stress Disorder in Patients Hospitalized With Traumatic Injuries. J Trauma Stress. 2021 Feb;34(1):104-115. doi: 10.1002/jts.22580. Epub 2020 Aug 17. PMID 33269808